CLINICAL TRIAL: NCT06375928
Title: Endoscopic Ultrasound-Guided Biliary Drainage With Lumen-Apposing Stent vs Classical ERCP for First-line Therapy of Malignant Distal Biliary Obstruction in Resectable Disease: An Open-label, Multicenter Randomized Controlled Trial (CARPEDIEM-1 Trial)
Brief Title: EUS-guided Choledochoduodenostomy vs ERCP as First Line in Malignant Distal Obstruction in Resectable Disease (CARPEDIEM-1 Trial)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari de Bellvitge (Other)
Collaborators: Hospital Mutua de Terrassa (Other); Hospital Clínico Universitario de Valencia (Other); Hospital General Universitario de Alicante (Other); Hospital Universitario Ramon y Cajal (Other); Hospital General Universitario de Castellón (Other); Hospital Álvaro Cunqueiro (Other); Complejo Hospitalario Universitario de Santiago (Other); University Hospital Virgen de las Nieves (Other); Complejo Hospitalario de Navarra (Other); Hospital de Sant Pau (Other); University of Salamanca (Other)
Responsible Party: Principal Investigator, Joan B Gornals, PhD and Head of Interventional Endoscopy Unit, Hospital Universitari de Bellvitge
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CARPEDIEM-1
Record Dates: First submitted 2024-04-16; First posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2023-08

CONDITIONS: Malignant Biliary Obstruction; Pancreatic Cancer Resectable; Biliary Tract Neoplasms
Keywords: Choledochoduodenostomy; Therapeutic endoscopy; Biliary Drainage; Lumen apposing metal stent; ERCP; Biliopancreatic maliognancy
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Self Expandable Metallic Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- ERCP with SEMS (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) with deployment of a self-expandable metallic stent (SEMS). Gold standard in malignant distal biliary obstruction (MDBO) in current practice.
  ERCP technique: Cannulation with papillotome (advanced cannulation techniques are allowed). Sphincterotomy. Self-expandable metallic stent (SEMS) deployment.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Self-expandable metallic stent (SEMS)
- EUS-CDS with LAMS-Pigtail (Experimental): Echoendoscopy-guided Choledochoduodenostomy (EUS-CDS) with deployment of a lumen-apposing metal stent (LAMS) and axis-orienting double-pigtail plastic stent throug LAMS.
  EUS-CDS technique: Diagnostic EUS. Classic or free-hand with preloaded guidewire choledochoduodenostomy with LAMS. Pneumatic dilation whithin LAMS is allowed. In case of bile duct < 15mm is mandatory the 'push' technique. Deployment of a pigtail coaxial to LAMS.
  Interventions: Procedure: Endoscopic biliary drainage; Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS)

INTERVENTIONS:
Procedure: Endoscopic biliary drainage — Decompression of the bile duct by endoscopic aproach.
  Other Names: Biliary drainage
Device: Self-expandable metallic stent (SEMS) — Self-expandable metallic stent (SEMS) deployment:
  * Covering: Uncovered or Partially Covered. Non covered if gallbladder is present.
  * Size: 10x40mm or 10x60mm or 10x80mm.
  Arms: ERCP with SEMS
Device: Lumen-apposing metal stent (LAMS) and double-pigtail plastic stent (DPPS) — Lumen-apposing metal stent (LAMS) with coaxial double-pigtail plastic stent (DPPS) deployment:
  * LAMS size: 6x8mm or 8x8mm. Consider 10x10mm if bile duct > 18mm.
  * DPPS size: 7Fr x 3-7cm.
  Arms: EUS-CDS with LAMS-Pigtail

SUMMARY:
The aim of this clinical trial is to evaluate temporal delay (days) between biliary drainage (EUS-CDS vs ERCP as first line therapy) and surgery in patients with resectable distal malignant biliary obstruction.

DETAILED DESCRIPTION:
Ecoendoscopy-guided choledochoduodenostomy (EUS-CDS) has been extended as a second line treatment in cases of ERCP failure in malignant distal biliary obstruction (MDBO). However, there are clinical trials which have compared it with ERCP as a first line treatment for MDBO in palliative patients, showing similar clinical and technical success and adverse events (AEs) rate between both techniques. Data about the benefit of this techique in resectable patients is still limited.

A recent retrospective study (Janet J et al, Ann Surg Oncol 2023) which included resectable patients, found that EUS-CDS group had significantly less delay (days) between biliary drainage and surgery than the ERCP group, with fewer endoscopy and surgery AEs.

Thus, our hypothesis is that EUS-CDS has benefits in terms of decreasing delay between biliary drainage when compared to ERCP in MDBO in resectable patients.

ELIGIBILITY:
Inclusion Criteria:

* Malignant distal biliary obstruction diagnosed in patient considered RESECTABLE with biliary drainage indication: i) impaired hepatic enzymes (including hyperbilirubinemia) x3 times upper the superior normal value. ii) Radiologic singns of extrahepatic bile duct obstruction with presence of retrograde dilatation, of at least 12-mm axial diameter.
* Consensual malignancy by a bilio-pancreatic multidisciplinar committe (histological confirmation is not mandatory)
* Patient capable of understanding and/or singning the informed consent.
* Patient who understands the type of study and will comply with all follow-up tests throughout its duration

Exclusion Criteria:

* Pregnancy or lactation.
* Severe coagulation disorder: INR > 1.5 non correctable with plasma administration and/or platelet count < 50.000/mm3.
* Distal malignant biliary strictures in patients considered borderline, non-surgical, unresectable, or palliative
* Benign or uncertain etiology of biliary strictures or strictures located proximally or in close proximity to the hilum.
* Patients with prior biliary stents or other biliary drainages (e.g., PTCD).
* Altered intestinal anatomy due to prior surgery that prevents or hinders papillary access (e.g., gastric bypass, Billroth II, duodenal switch, Roux-en-Y).
* Stenosis in the antral or duodenal region that prevents access to the duodenum and reaching the papilla.
* Situations that do not allow for upper gastrointestinal endoscopy (e.g., esophageal stricture).
* Patients with functional diversity, who lack the capacity to understand the nature and potential consequences of the study, except when a legal representative is available.
* Patients incapable of maintaining follow-up appointments (lack of adherence).
* Lack of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Delay in days between endoscopic biliary drainage and cephalic duodenopancreatectomy (CDP) | 1 day to 12 months
  Number of days between intervention (T1-biliary drainage) and surgery.

SECONDARY OUTCOMES:
Technical success | day 0
  ERCP group: cannulation, cholangiogram, correct deployment of SEMS. EUS-CDS group: Correct deployment of both flaps of LAMS (and pigtail) in place, checked by ecoendoscopy/endoscopic image/floroscopy.
Clinical success | 14 days after BD
  In jaundice: decreasing > 50% of bilirrubin or normalization of bilirrubin levels 14 days after endoscopic procedure.
  In cholangitis: stop of antibiotics without clinical recurrence or decreasing > 50% of acute phase reactants 14 days after the endoscopic procedure.
AE - biliary drainage | 0 to 30 days after BD
  Adverse events rate related to biliary drainage according to the AGREE classification
AE - surgery | 0 to 90 days after surgery
  Adverse events rate related to surgery according to the Claiven and Dindo classification.

CONTACTS AND LOCATIONS:
Overall Officials: Joan B Gornals, PhD, Principal Investigator — Bellvitge University Hospital
Locations (1):
- Hospital Universitari de Bellvitge, L'Hospitalet de Llobregat, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Teoh AYB, Napoleon B, Kunda R, Arcidiacono PG, Kongkam P, Larghi A, Van der Merwe S, Jacques J, Legros R, Thawee RE, Saxena P, Aerts M, Archibugi L, Chan SM, Fumex F, Kaffes AJ, Ma MTW, Messaoudi N, Rizzatti G, Ng KKC, Ng EKW, Chiu PWY. EUS-Guided Choledocho-duodenostomy Using Lumen Apposing Stent Versus ERCP With Covered Metallic Stents in Patients With Unresectable Malignant Distal Biliary Obstruction: A Multicenter Randomized Controlled Trial (DRA-MBO Trial). Gastroenterology. 2023 Aug;165(2):473-482.e2. doi: 10.1053/j.gastro.2023.04.016. Epub 2023 Apr 28. PMID 37121331
- [Result] Janet J, Albouys J, Napoleon B, Jacques J, Mathonnet M, Magne J, Fontaine M, de Ponthaud C, Durand Fontanier S, Bardet SSM, Bourdariat R, Sulpice L, Lesurtel M, Legros R, Truant S, Robin F, Prat F, Palazzo M, Schwarz L, Buc E, Sauvanet A, Gaujoux S, Taibi A. Pancreatoduodenectomy Following Preoperative Biliary Drainage Using Endoscopic Ultrasound-Guided Choledochoduodenostomy Versus a Transpapillary Stent: A Multicenter Comparative Cohort Study of the ACHBT-FRENCH-SFED Intergroup. Ann Surg Oncol. 2023 Aug;30(8):5036-5046. doi: 10.1245/s10434-023-13466-8. Epub 2023 Apr 17. PMID 37069476
- [Result] Paik WH, Lee TH, Park DH, Choi JH, Kim SO, Jang S, Kim DU, Shim JH, Song TJ, Lee SS, Seo DW, Lee SK, Kim MH. EUS-Guided Biliary Drainage Versus ERCP for the Primary Palliation of Malignant Biliary Obstruction: A Multicenter Randomized Clinical Trial. Am J Gastroenterol. 2018 Jul;113(7):987-997. doi: 10.1038/s41395-018-0122-8. Epub 2018 Jul 2. PMID 29961772
- [Result] Bang JY, Hawes R, Varadarajulu S. Endoscopic biliary drainage for malignant distal biliary obstruction: Which is better - endoscopic retrograde cholangiopancreatography or endoscopic ultrasound? Dig Endosc. 2022 Jan;34(2):317-324. doi: 10.1111/den.14186. Epub 2021 Nov 29. PMID 34748675